CLINICAL TRIAL: NCT01970202
Title: Comparing the Efficacy of Two Frequently Used Doses of Enoxaparin for VTE Prophylaxis After Bariatric Surgery
Brief Title: Anti Xa Levels Under Two Different Regimens of Enoxaparin VTE Prophylaxis After Sleeve Gastrectomy for Morbid Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Nachum vaisman, Prof, Principle investigator, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-13-GL-0241-CTIL
Record Dates: First submitted 2013-10-14; First posted 2013-10-28 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Obesity
Keywords: obesity; overweight; sleeve gastrectomy
MeSH Terms: conditions — Obesity; Overweight | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40mg Enoxaparin (Active Comparator): Patients with obesity undergoing laparoscopic sleeve gastrectomy, will receive 40mg Enoxaparin per day for 3 days after surgery by subcutaneous administration.
  Interventions: Drug: 40mg Enoxaparin
- 60mg Enoxaparin (Active Comparator): Patients with obesity undergoing laparoscopic sleeve gastrectomy, will receive 60mg Enoxaparin per day for 3 days after surgery by subcutaneous administration.
  Interventions: Drug: 60mg Enoxaparin
- Control (Other): no treatment
  Interventions: Other: Control

INTERVENTIONS:
Drug: 40mg Enoxaparin — Patients with obesity undergoing laparoscopic sleeve gastrectomy, will receive 40mg Enoxaparin per day for 3 days after surgery by subcutaneous administration.
  Other Names: clexane
  Arms: 40mg Enoxaparin
Drug: 60mg Enoxaparin — Patients with obesity undergoing laparoscopic sleeve gastrectomy, will receive 60mg Enoxaparin per day for 3 days after surgery by subcutaneous administration.
  Other Names: clexane
  Arms: 60mg Enoxaparin
Other: Control — no treatment
  Arms: Control

SUMMARY:
Approximately two thirds of the adult population in developed countries is categorized as over-weight or obese (BMI>30). In spite of worldwide increasing awareness, obesity is a major health concern. In the presence of numerous diets, medical therapies, and robust research, bariatric surgery remains the most effective means of weight reduction in morbidly obese patients (BMI>40, or BMI>35 with co-morbidities). However, bariatric surgery harbors a relatively high risk for postoperative complications; of them, venous thromboembolic events (VTE) are not common, but potentially lethal. Taken together with the propensity of morbidly obese patients to develop VTE, perioperative thromboprophylaxis is mandatory.

To date, low molecular weight heparins (LMWH) are most commonly used for VTE prophylaxis in the aforementioned population. Due to the pharmacologic properties of LMWH and the characteristics of surgically treated obese patients, the optimal dose that is to be utilized for VTE prophylaxis in this population remains unclear. Assessment of anti-FXa levels in the patients' plasma can be used in order to monitor LMWH activity. Levels of 0.2-0.5 U/ml have been proposed by some authors for VTE prophylaxis.

Few studies have compared different dosing regimens of enoxaparin (between 30mg-60mg q/12h) for VTE prophylaxis in the population undergoing bariatric surgery; nevertheless, these were small non- randomized trials, containing numerous methodological weaknesses. Hence, the optimal regimen of enoxaparin to be used for the prevention of VTE in the discussed population remains unclear.

The aim of the present study is to evaluate plasma levels of anti-FXa activity, comparing two most commonly used enoxaparin prophylactic regimens (40mg vs 60mg q/24h) in a large and homogenous cohort of sleeve gastrectomy patients. Although universally used by bariatric surgeons, the pharmacologic efficacy of these regimens has not been evaluated in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
The following steps shall be performed in the process of recruiting a patient for the study:

Preoperatively:

* A baseline blood sample for Anti-FXa levels shall be obtained.
* Randomization of the patient to one of the two treatment groups

Postoperatively:

* All patients will be treated with Sequential Compression Devices, massive I.V hydration and encouraged to ambulate early.
* Patients will receive three injections of enoxaparin, according to the treatment group they were assigned to, The first injection given on the morning after surgery. Four hours after the third injection of enoxaparin a blood sample will be taken from the patients and assessed for anti-FXa levels.

A control group of 5 patients, randomly elected, will be recruited. This group will not be treated with enoxaparin. These patients will be treated with sequential compression devices and massive I.V hydration, an accepted treatment, proven effective for the studied population. The goal is to assess the anti-FXa levels in these patients, representing the baseline levels in patients undergoing laparoscopic sleeve gastrectomy.

Furthermore, the preoperative, operative and postoperative management of these patients will be identical to that of the treatment groups and on the third day post-operation a blood sample from these patients will be retrieved and assessed for anti-FXa levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing laparoscopic sleeve gastrectomy.
* The patient undergoes the surgery in the surgical wing of the Tel-Aviv Sourasky Medical Center.
* The patient has received full information regarding the studies nature, has agreed to participate and has given informed consent (documented by a signed informed consent form).

Exclusion Criteria:

* Patients with a previous Venous Thromboembolic Event.
* Patients requiring an IVC filter.
* Patients with known thrombophilia due to coagulation factor disorders (i.e factor V leiden).
* Patients with a bleeding disorder
* Patients with renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Anti-factor Xa plasma levels | within 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guy Lahat, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel

REFERENCES:
- [Derived] Amaral FC, Baptista-Silva JC, Nakano LC, Flumignan RL. Pharmacological interventions for preventing venous thromboembolism in people undergoing bariatric surgery. Cochrane Database Syst Rev. 2022 Nov 22;11(11):CD013683. doi: 10.1002/14651858.CD013683.pub2. PMID 36413425